CLINICAL TRIAL: NCT02466412
Title: A Single-center, Open-label, Randomized, Controlled, Crossover Study to Investigate the Nicotine Pharmacokinetic Profile of the Carbon Heated Tobacco Product 1.1 Menthol (CHTP 1.1 M) Following Single Use in Smoking, Healthy Subjects Compared to Menthol Conventional Cigarettes
Brief Title: Nicotine Pharmacokinetic Profile of the CHTP 1.1 M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P2M-PK-04-JP; P2M-PK-04-JP (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2015-05-07; First posted 2015-06-09 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Smoking
Keywords: smoking; nicotine absorption; potential modified risk tobacco product; cigarette; Carbon Heated Tobacco Product
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHTP 1.1 M then mCC (Active Comparator): Each subject will follow the below study design:
  * Day -1 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of CHTP 1.1 M)
  * Day 2 = Wash-out
  * Day 3 = 2nd intervention (single product use of mCC).
  Interventions: Other: CHTP 1.1 M; Other: mCC
- mCC then CHTP 1.1 M (Active Comparator): Each subject will follow the below study design:
  * Day -1 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of mCC)
  * Day 2 = Wash-out
  * Day 3 = 2nd intervention (single product use of CHTP 1.1 M).
  Interventions: Other: CHTP 1.1 M; Other: mCC

INTERVENTIONS:
Other: CHTP 1.1 M — Single use of the Carbon Heated Tobacco Product 1.1 Menthol (CHTP 1.1 M)
Other: mCC — Single use of subject's own menthol conventional cigarette (mCC)

SUMMARY:
The primary objective of this clinical study is to evaluate the pharmacokinetic (PK) profile of nicotine (rate and amount of nicotine absorbed) after single use of the Carbon Heated Tobacco Product 1.1 Menthol (CHTP 1.1 M), a potential Modified Risk Tobacco Product, compared to menthol cigarettes (mCC) in healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese.
* Subject is at a minimum 23 years of age.
* Smoking, healthy subject as judged by the Investigator.
* Subject has smoked for at least the last 3 years
* Subject smoked at least 10 commercially available mCCs per day over the last 4 weeks.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of a drug (whichever is longer) which has an impact on CYP2A6 activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Fumimasa Nobuoka, MD, Principal Investigator — Ageo Medical Clinic
Locations (1):
- Ageo Medical Clinic, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 08 May 2015
  On Day -3 (admission), after all inclusion/exclusion criteria were checked, all eligible subjects were enrolled and tried CHTP 1.1 M.
  From enrollment, they were asked to remain abstinent from smoking for at least 24 hours before being randomized on Day 1 into 1 of the 2 sequences.
Pre-assignment Details: Number of subjects enrolled = 56, but only 48 were randomized as described below:
  * Sequence "CHTP 1.1 M then mCC": 24 subjects
  * Sequence "mCC then CHTP 1.1 M": 24 subjects
  Number of subjects enrolled but NOT randomized = 8
Period: Washout Period of 1 Day (Day -1)
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: First Intervention (Day 1)
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Washout Period of 1 Day (Day 2)
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Second Intervention (Day 3)
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall PK population consisted of 47 subjects.
  1 subject was excluded from the PK population (sequence "CHTP 1.1 M then mCC" ) due to all plasma nicotine concentration measurements being below the quantification limit for both CHTP 1.1 M and mCC.
Groups:
- Total: Total of all reporting groups
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (10.03) | 40.7 (11.48) | 42.6 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 12 | 10 | 22
International Organization for Standardization (ISO) nicotine Yield [Count of Participants; unit: Participants]
  ≤ 0.6 mg | 11 | 11 | 22
  > 0.6 to ≤ 1 mg | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of CHTP 1.1 M and mCC
Description: T0 = start of single product use.
  Derived from multiple blood sampling on Day 1 and Day 3 (1 blood sampling pre-product use and multiple blood sampling over 24 hours post-product use).
  Geometric Least Squares (LS) means are provided.
Time Frame: Day 3: blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0.
Population: The PK population consisted of 47 subjects.
  1 subject was excluded from the PK population (sequence "CHTP 1.1 M then mCC") due to all plasma nicotine concentration measurements being below the quantification limit for both CHTP 1.1 M and mCC.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- CHTP 1.1 M: The geometric least square mean presented below takes into consideration the data of all the subjects included in the PK population after single use of CHTP 1.1 M.
- Menthol Cigarette (mCC): The geometric least square mean presented below takes into consideration the data of all the subjects included in the PK population after single use of mCC.
Arm/Group | CHTP 1.1 M | Menthol Cigarette (mCC)
Number analyzed (Participants) | 47 | 47
ng/mL | 6.2950 [5.2610 to 7.5322] | 9.8463 [8.2290 to 11.7815]
Statistical Analysis 1: Comparison: CHTP 1.1 M vs Menthol Cigarette (mCC); The objective of this study was to determine the point estimate and precision of the CHTP 1.1 M:mCC ratio for Cmax. Therefore, there was no statistical hypothesis to be tested for this objective; Test type: Superiority or Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 63.9326, 95% CI 2-sided [49.6045 to 82.3991] — Geometric LS mean ratio (CHTP 1.1 M:mCC). Expressed as %

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero (Pre-product Use) to Last Time Point [AUC(0-last)] Following Single Use of CHTP 1.1 M and mCC
Description: T0 = start of single product use.
  Derived from multiple blood sampling on Day 1 and Day 3 (1 blood sampling pre-product use and multiple blood sampling over 24 hours post-product use).
  Geometric Least Squares means are provided.
Time Frame: Day 3: blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | CHTP 1.1 M | Menthol Cigarette (mCC)
Number analyzed (Participants) | 47 | 47
h*ng/mL | 8.5311 [6.9550 to 10.4642] | 14.2172 [11.5908 to 17.4388]
Statistical Analysis 1: Comparison: CHTP 1.1 M vs Menthol Cigarette (mCC); The objective of this study was to determine the point estimate and precision of the CHTP 1.1 M:mCC ratio for AUC(0-last). Therefore, there was no statistical hypothesis to be tested for this objective; Test type: Superiority or Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 60.0052, 95% CI 2-sided [44.9517 to 80.0997] — Geometric LS mean ratio (CHTP 1.1 M:mCC). Expressed as %

ADVERSE EVENTS:
Time Frame: From the informed consent form (ICF) signature until the end of the safety follow-up period (7 days after discharge of the subject).
Description: The safety was assessed in the safety population, consisting of 56 subjects: 48 randomized subjects (24 subjects in the "CHTP 1.1 M then mCC" sequence, 24 subjects in the "mCC then CHTP 1.1 M" sequence), and 8 non-randomized subjects who were exposed to CHTP 1.1 M from the product test on Admission.
Groups:
- Enrolled But Not Randomized: Subjects who tried the CHTP 1.1 M at Admission but were not randomized in 1 of the 2 sequences as they were back-up subjects
Arm/Group | CHTP 1.1 M Then mCC | mCC Then CHTP 1.1 M | Enrolled But Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/8
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02466412/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02466412/SAP_001.pdf